CLINICAL TRIAL: NCT00604357
Title: A Pilot Study to Determine the Safety and Efficacy of Induction-Therapy, De Novo MPA and Delayed mTOR-Inhibition in Liver Transplant Recipients With Impaired Renal Function. (PATRON-Study)
Brief Title: CNI-free de Novo Protocol in Patients Undergoing Liver Transplantation With Renal Impairment
Acronym: PATRON07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Hans J Schlitt, Prof. MD, Professor Dr. Hans J Schlitt, University of Regensburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PATRON07
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: End Stage Liver Disease; Impaired Renal Function
Keywords: CNI free; mTOR inhibition; induction; IL2 receptor antibodies; renal function; liver transplantation
MeSH Terms: conditions — End Stage Liver Disease; Renal Insufficiency | interventions — Sirolimus; Basiliximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Prior to reperfusion 500 mg Prednisolone will be administered i.v.. After the transplantation, a combination of anti-CD25-mAB (basiliximab 20 mg on day 0 and day 4 after the procedure), and MMF 2 g/d, 2 applications per day i.v., later conversion to oral intake) will be applied. Earliest, on day 10 after LT Sirolimus will be introduced aiming at 24 hours trough-levels for Sirolimus between 4 and 8 ng/mL. Steroids will be started on day 1 after transplantation with 1mg/kg BW and will be tapered every 2 days for 5 mg to a dosage of 20 mg and for 2.5 mg every two days to 7.5 mg. Thereafter the dosage will be reduced to 5 mg and 2.5 mg for 1 week each and eliminated thereafter. Additionally, every patient with risk constellation will receive cytomegalovirus (CMV) prophylaxis and prophylaxis against Pneumocystis carinii infection during the first 3 months after liver transplantation.
  Interventions: Drug: anti-CD 25 mAb, Sirolimus, MMF

INTERVENTIONS:
Drug: anti-CD 25 mAb, Sirolimus, MMF — Prior to reperfusion: 500 mg Prednisolone After OLT: anti-CD25-mAB (basiliximab 20 mg on day 0 and day 4 after the procedure)
  MMF 2 g/d, 2 applications per day i.v., later conversion to oral intake)
  Earliest, on day 10 after LT Sirolimus: 5 mg/d, thereafter a dosage of 2 mg/d (4 and 8 ng/mL)
  Steroids: 1mg/kg BW (tapered every 2 days for 5 mg to a dosage of 20 mg, 2.5 mg every two days to 7.5 mg, reduced to 5 mg and 2.5 mg for 1 week each and eliminated thereafter).
  Other Names: Rapamune; Simulect; CellCept; DecortinH

SUMMARY:
Background:

Patients undergoing liver transplantation with preexisting renal dysfunction are prone to further renal impairment with the early postoperative use of Calcineurin-inhibitors. However, there is only little scientific evidence for the safety and efficacy of de novo CNI free regimens in patients with impaired renal function undergoing liver transplantation. The objective of the study is to evaluate a de novo calcineurin-inhibitor-free immunosuppressive regimen based on induction therapy with anti-CD25 monoclonal anti- body, mycophenolate mofetil (MMF/MPA), and mTOR-inhibition to determine its safety and to investigate the preliminary efficacy in patients with impaired renal function at the time of liver transplantation. Methods/Design: Patients older than 18 years with renal impairment at the time of liver transplantation due to hepatorenal syndrome, eGFR < 50 ml/min and/or serum creatinine levels > 1.5 mg/dL will be included. Patients will receive a combination therapy with antiCD25-monoclonal antibodies, MMF, steroids and delayed sirolimus (day 10) and will be evaluated with regards to the incidence of steroid resistant acute rejection within the first 30 days after liver transplantation as the primary endpoint. The study is designed as prospective two-step trial requiring a maximum of 29 patients. In the first step 9 patients will be included. If 8 or more patients show no signs of biopsy proven steroid resistant rejection, additional 20 patients will be included. If in the second step a total of 27 or more patients reach the primary end-point the regimen is regarded to be safe and efficient. The follow up period will be one year after transplantation. The aim is to obtain safety and efficacy data for this new and innovative therapy regimen that might be the basis for a large prospective randomized multicenter trial in the future.

DETAILED DESCRIPTION:
Objectives of this study The objective of the study is to evaluate a de novo CNI-free immunosuppressive regimen based on induction therapy with anti-CD25 monoclonal anti- body, mycophenolate mofetil (MMF/MPA), and delayed mTOR-inhibition. The primary endpoint is defined as the incidence of steroid-resistant acute rejection within the first 30 days after liver transplantation.

Secondary objectives include the incidence of acute rejection(s), the number and the timing of acute rejections per patient within the first year after transplantation. A critical secondary endpoint will be the development of renal function at 1 week, 1, 3, 6 and 12 months after liver transplantation. This includes information on the number of patients requiring renal replacement therapy and its duration. During follow-up of 1 year liver allograft function, infectious complications, treatment failures defined as introduction of CNIs as well as side-effects affecting the hematopoetic system, tolerability, impaired wound-healing, the incidence of hepatic artery thrombosis and mortality will be explicitly documented and investigated.

Trial population The collective we are aiming at are patients older than 18 years with a preexisting renal impairment at the time of liver transplantation. Patients will be eligible if the eGFR < 50 ml/min (Cockcroft-Gault) and/or their serum creatinine levels > 1.5 mg/dL.

Follow-Up Every patient will be followed up for 1 year after transplantation. The primary end-point will be at 30 days after transplantation (Steroid resistant acute rejection). During the first 30 days after transplantation there will be 9 visits where laboratory values (liver, renal and metabolic function, sirolimus trough levels), adverse events and rejection episodes will be recorded. Additionally there will be an ultrasound on day 1 after liver transplantation and on day 10 prior to the initiation of sirolimus to exclude hepatic artery thrombosis.

Between day 30 and 1 year after liver transplantation the patient will be followed up to evaluate the long time outcome and secondary objectives of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary liver transplantation.
* Patients older than 18 years.
* Patients with a hepatorenal syndrome type I or II
* eGFR < 50 ml/min at the time point of transplantation
* Serum creatinine levels > 1.5 mg/dL at the time-point of transplantation

Exclusion Criteria:

* Patients with pre-transplant renal replacement therapy > 14 days.
* Patients with a known hypersensitivity to mTOR-inhibitors.
* Patients with a known hypersensitivity to mycophenolate acid.
* Patients with a known hypersensitivity to anti CD 25-monoclonal antibodies.
* Patients with platelets < 50.000/nl.
* Patients with triglycerides > 350 mg/dl and cholesterol > 300 mg/dl refractory to optimal medical treatment prior to initiation of therapy with mTOR inhibition.
* Severe systemic infections and wound-healing disturbances prior to inclusion.
* Multiple organ graft recipients.
* Patients with signs of a hepatic artery stenosis directly prior to initiation of therapy with Sirolimus.
* Patients with a psychological, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule.
* Patients under guardianship (e.g. individuals who are not able to freely give their informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined as the incidence of steroid-resistant acute rejection within the first 30 days after liver transplantation. | 30 days

SECONDARY OUTCOMES:
incidence of acute rejection(s) | 1 year
the number and the timing of acute rejections | 1 year
the development of renal function at 1 week, 1, 3, 6 and 12 months after liver transplantation | 1 year
liver allograft function | 1 year
infectious complications | yes
treatment failures defined as introduction of CNIs | 1 year
side-effects affecting the hematopoetic system | 1 year
tolerability | 1 year
impaired wound-healing | 1 year
incidence of hepatic artery thrombosis | 1 year
mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas A Schnitzbauer, MD, Study Director — Regensburg University Medical Center, Department of Surgery; Hans J Schlitt, MD, Study Chair — Regensburg University Medical Center, Department of Surgery; Marcus N Scherer, MD, Principal Investigator — Regensburg University Medical Center, Department of Surgery
Locations (1):
- Regensburg University Medical Center, Department of Surgery, Regensburg, Bavaria, Germany

REFERENCES:
- [Derived] Schnitzbauer AA, Sothmann J, Baier L, Bein T, Geissler EK, Scherer MN, Schlitt HJ. Calcineurin Inhibitor Free De Novo Immunosuppression in Liver Transplant Recipients With Pretransplant Renal Impairment: Results of a Pilot Study (PATRON07). Transplantation. 2015 Dec;99(12):2565-75. doi: 10.1097/TP.0000000000000779. PMID 26018348
- [Derived] Schnitzbauer AA, Scherer MN, Rochon J, Sothmann J, Farkas SA, Loss M, Geissler EK, Obed A, Schlitt HJ. Study protocol: a pilot study to determine the safety and efficacy of induction-therapy, de novo MPA and delayed mTOR-inhibition in liver transplant recipients with impaired renal function. PATRON-study. BMC Nephrol. 2010 Sep 14;11:24. doi: 10.1186/1471-2369-11-24. PMID 20840760